CLINICAL TRIAL: NCT05900518
Title: A Promising Minimally Invasive Surgical Technique for the Treatment of Infected Pilonidal Sinus
Acronym: LASER SILAT
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: LASER SILAT
Record Dates: First submitted 2023-05-31; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Infected Pilonidal Sinus
Keywords: laser

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Infected pilonidal sinuses are a common pathology, affecting an estimated 0.7% of the population. In France, the most commun technique is extended exeresis with an open wound, followed by directed healing. This technique reduces the risk of recurrence, albeit at the cost of daily nursing care and a long healing period involving prolonged absence from work. Closure or plasty surgical techniques aimed at reducing the duration of nursing care are more restrictive, and seem to have higher recurrence rate. Minimally invasive treatment, such as phenolization and flattening with curettage of the sinus have existed for over 50 years, albeit with disappointing long-term results and morbidity that limits their application.

Today, new minimally invasive treatments are being developed, aiming at a less constraining post-operative period. without compromising healing. These include glue, endoscopic treatment (EPSiT : Endoscopic Pilonidal Sinus Treatment or VAASP : Video-Assisted Ablation of Pilonidal Sinus) and laser treatment (SiLaT procedure : Sinus Laser Therapy or PiLaT : Pilonidal disease Laser Treatment).

Laser treatment is used since 2014 in the treatment of anal fistulas and more recently in the treatment of infected pilonidal sinus. A laser fiber is introduced, under local or general anaesthesia, into the main cavity and secondary tracts after curettage and opening of the dimples. The energy delivered by the laser is transmitted in the form of heat, in order to seal the cavity during healing of thermal lesions.

Initial results report success rates of around 90%, with a healing time of between 1 and 2 months. It also appears to be effective after failure of previous surgery. In cases of incomplete closure or recurrence, a second laser treatment can be performed with high healing rates. The investigators carried out an retrospective study including 29 patients treated with the SILAT technique. The healing rate, defined as the absence of symptoms and recurrence of suppuration, was around 70%. The procedure was painless and no serious complications were observed. The presence of one or more secondary orifices and overweight were associated with a higher risk of failure.

In order to confirm these results, to better specify the factors predictive of success, and to evaluate the efficacy of SiLaT in the longer term, the investigators will carry out a single-center study including all adult patients treated with laser between June 2018 and December 2020.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 or above
* French-speaking patient
* Patient hospitalized in the Proctology department of GHPSJ between 01JUN2018 and 31DEC2020 for a chronically infected pilonidal sinus
* patient presenting an recurring infected pilonidal sinus after open or closed surgical treatment

Exclusion Criteria:

* Patient hospitalized in the acute abcess stage of an infected pilonidal sinus
* Patient under guardianship or curatorship
* Patient incarcerated
* Patient under legal protection
* Patient refusing enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient hospitalized in the Proctology department of GHPSJ between 01JUN2018 and 31DEC2020 for a chronically infected pilonidal sinus
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2021-10-14 (Actual)

PRIMARY OUTCOMES:
Clinical cure | between 6 months and 36 months after treatment
  A clinical evaluation will be performed and Clinical cure will be defined by : closure of all existing fistula external opening AND absence of abscess, AND absence of leakage under pressure, and ABSENCE of pain

SECONDARY OUTCOMES:
recurrence Rate | between 6 months and 36 months after treatment
  number of recurrence in the study population
Incidence rate of complication after laser treatment | between 6 months and 36 months after treatment
  incidence rate of fever, abcess, acute urinary retention, bleeding or other complication
description of predictive failure factors | between 6 months and 36 months after treatment
  incidence rate of smoking habits, diabetes, inflammatory bowel disease, anal fistula, Verneuil disease, other proctological disease, previous surgery for the infected pilonidal disease among the relapsing patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Parades V, Bouchard D, Janier M, Berger A. Pilonidal sinus disease. J Visc Surg. 2013 Sep;150(4):237-47. doi: 10.1016/j.jviscsurg.2013.05.006. Epub 2013 Aug 1. PMID 23911903
- [Background] Johnson EK, Vogel JD, Cowan ML, Feingold DL, Steele SR; Clinical Practice Guidelines Committee of the American Society of Colon and Rectal Surgeons. The American Society of Colon and Rectal Surgeons' Clinical Practice Guidelines for the Management of Pilonidal Disease. Dis Colon Rectum. 2019 Feb;62(2):146-157. doi: 10.1097/DCR.0000000000001237. No abstract available. PMID 30640830
- [Background] Pappas AF, Christodoulou DK. A new minimally invasive treatment of pilonidal sinus disease with the use of a diode laser: a prospective large series of patients. Colorectal Dis. 2018 Aug;20(8):O207-O214. doi: 10.1111/codi.14285. Epub 2018 Jun 27. PMID 29878584
- [Background] Georgiou GK. Outpatient laser treatment of primary pilonidal disease : the PiLaT technique. Tech Coloproctol. 2018 Oct;22(10):773-778. doi: 10.1007/s10151-018-1863-5. Epub 2018 Oct 10. PMID 30306277
- [Background] Dessily M, Charara F, Ralea S, Alle JL. Pilonidal sinus destruction with a radial laser probe: technique and first Belgian experience. Acta Chir Belg. 2017 Jun;117(3):164-168. doi: 10.1080/00015458.2016.1272285. Epub 2017 Jan 6. PMID 28056720